CLINICAL TRIAL: NCT01334164
Title: Recovery Management Checkups for Women Offenders Experiment
Brief Title: Recovery Management Checkups for Women Offenders
Acronym: RMC-WO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: Haymarket Center (Other); Cook County Sheriff's Women's Justice Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1037-0905; R01DA021174 (NIH)
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Recovery Management Checkup (RMC); Outcome Monitoring
Keywords: substance use disorder; offenders; reentry; HIV risk behavior; recidivism
MeSH Terms: conditions — Substance-Related Disorders; Recidivism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recovery Management Checkup (RMC) (Experimental): Women assigned to the RMC condition met with a linkage manager after each research interview. When a woman reported substance use, HIV risk behavior or illegal activity, the linkage manager used motivational interviewing to: provide feedback regarding her current substance use, HIV risk behavior or illegal activity, discuss barriers that prevented her from stopping each activity and ways of avoiding them in the future, and assess and discuss her level of motivation for change. Linkage managers also scheduled treatment appointments, accompanied the women to treatment intake and stayed through the process and implemented an Engagement and Retention Protocol designed to improve retention rates. For women who refused the treatment option, the linkage manager and participant agreed upon an Alternative Action plan, which included various behaviors the woman had agreed to engage in to reduce or stop her substance use, HIV risk, or her participation in illegal activity.
  Interventions: Behavioral: Recovery Management Checkups
- Outcome Monitoring (Active Comparator): Outcome monitoring only, however participates are still able (and do) enter treatment on their own.
  Interventions: Other: Outcome Monitoring

INTERVENTIONS:
Behavioral: Recovery Management Checkups — Women assigned to the RMC condition met with a linkage manager after each research interview. When a woman reported substance use, HIV risk behavior or illegal activity, the linkage manager used motivational interviewing to: provide feedback regarding her current substance use, HIV risk behavior or illegal activity, discuss barriers that prevented her from stopping each activity and ways of avoiding them in the future, and assess and discuss her level of motivation for change. Linkage managers also scheduled treatment appointments, accompanied the women to treatment intake and stayed through the process and implemented an Engagement and Retention Protocol designed to improve retention rates. For women who refused the treatment option, the linkage manager and participant agreed upon an Alternative Action plan, which included various behaviors the woman had agreed to engage in to reduce or stop her substance use, HIV risk, or her participation in illegal activity.
  Arms: Recovery Management Checkup (RMC)
Other: Outcome Monitoring — Outcome monitoring only, however participates are still able (and do) enter treatment on their own
  Arms: Outcome Monitoring

SUMMARY:
The proposed study is designed to test the effectiveness of recovery management checkups for women offenders (RMC-WO) released from jail to provide continuity of care immediately upon release and to help them manage their long-term recovery. The hypotheses in the first phase were: 1)women assigned to RMC (versus control) will a) return to treatment sooner after the initial release from jail and b) be more likely to receive treatment in the 90 days after release from jail; 2)women who received treatment in the first 90 days post release (vs. no treatment) will be more likely to sustain their abstinence through 90 days post release from a) any alcohol or drugs, b) alcohol, c) cannabis, d) cocaine, and e) opiates; 3)women who maintained their abstinence from any alcohol and other drugs through the first 90 days post release (vs. any relapse) will be less likely to have a) unprotected sex, b) commit any other illegal activity, and d) be re-incarcerated in jail or prison. In the second phase repeated exposure to these efforts on a quarterly basis is expected to further strengthen each of these effects.

DETAILED DESCRIPTION:
The components of the recovery management checkups will include: on-going monitoring via a re-entry meeting, two monthly meetings and quarterly assessments for 3 years, personalized feedback on substance use and high risk behaviors, linkage to community-based substance abuse treatment (when needed), on-site HIV booster sessions (when needed), and treatment engagement and retention support. Motivational interviewing will provide the therapeutic approach to transition women from one step of the change process to another. Combined, these components and therapeutic milieu afford an opportunity for immediate linkage to community-based treatment and HIV prevention as well as ongoing monitoring for relapse and early re-intervention for both substance use and HIV risk behaviors (both public health priorities).

ELIGIBILITY:
Phase 1

Inclusion Criteria:

* adult women offenders with substance problems re-entering the community from county jail programs

Exclusion Criteria:

* had not used substances in the 90 days before incarceration
* had no abuse/dependence symptoms
* were under 18 years old
* lived or planned to move outside Chicago within the next 12 months
* were not fluent in English or Spanish
* were cognitively unable to provide informed consent and were released before the 14th day of incarceration Phase 2

Inclusion Criteria:

* released to the community
* agreed to participate in the study
* completed the initial interview

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2007-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Time to treatment re-entry | 3 years post release
  Time from first relapse (after release from jail) to first treatment re-entry measured in days and censored at the last observation.
Any Treatment | Quarterly and over 3 years
  Receipt of any substance abuse treatment during each quarter and overall all observed quarters.

SECONDARY OUTCOMES:
Abstinence | Quarterly and over 3 years
  Based on no self reported use and clean urine tests at 30, 60 and 90 days post release for: a) any alcohol or drugs, b) alcohol, c) cannabis, d) cocaine, and e) opiates
HIV risk behaviors and Recidivism | Quarterly and over 3 years
  Based on no self report post release of a) unprotected sex defined as having vaginal, anal or oral sex without a barrier like a male condom, women's condom, or dental dam.; b) no self reported illegal activity other than drug use and no arrest; and c) no days in jail or prison.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chestnut Health Systems-Lighthouse Institute, Chicago, Illinois
  - Chestnut Health Systems, Normal, Illinois

REFERENCES:
- [Derived] Scott CK, Dennis ML. The first 90 days following release from jail: findings from the Recovery Management Checkups for Women Offenders (RMCWO) experiment. Drug Alcohol Depend. 2012 Sep 1;125(1-2):110-8. doi: 10.1016/j.drugalcdep.2012.03.025. Epub 2012 Apr 27. PMID 22542465